CLINICAL TRIAL: NCT06374433
Title: Investigating the Plasticity of Human Predictive Coding Through Neuromodulation: an Interventional, Monocentric, Randomized, Single-blinded Study on Healthy Adult Volunteers
Brief Title: Investigating the Plasticity of Human Predictive Coding Through Neuromodulation
Acronym: PREDICOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università Vita-Salute San Raffaele (Other)
Collaborators: Alessia Santoni (Unknown); Sara Stottmeier (Unknown); Klara Hemmerich (Unknown); Giuseppe Di Dona (Unknown); Luigi Ferini-Strambi (Unknown)
Responsible Party: Principal Investigator, Luca Ronconi, Professor, Università Vita-Salute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PREDICOM-01
Record Dates: First submitted 2024-04-08; First posted 2024-04-18 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Human Brain and Cognition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Occipital tACS at IAF-2Hz (Experimental): Transcranial alternating current stimulation (tACS) at occipital sites to modulate the occipital brain areas' activity at a frequency below the individual alpha frequency (IAF-2 Hz).
  Interventions: Procedure: Occipital tACS at IAF-2Hz
- Occipital tACS at IAF+2Hz (Experimental): Transcranial alternating current stimulation (tACS) at occipital sites to modulate the occipital brain areas' activity at a frequency above the individual alpha frequency (IAF+2 Hz).
  Interventions: Procedure: Occipital tACS at IAF+2Hz
- Frontal tACS at 4-7 Hz (Experimental): Transcranial alternating current stimulation (tACS) at frontal sites to modulate the frontal brain areas' activity at a frequency within the theta band (4-7 Hz).
  Interventions: Procedure: Frontal tACS at 4-7 Hz
- Sham/placebo tACS (Sham Comparator): Transcranial alternating current stimulation (tACS) is applied only in the first and the last 30 seconds of the experimental procedure, thus resulting ineffective.
  Interventions: Procedure: Sham/placebo tACS
- Occipital tRNS (Experimental): Stimulation at occipital sites with transcranial random noise stimulation (tRNS) to modulate occipital brain areas plasticity
  Interventions: Procedure: Occipital tRNS
- Frontal tRNS (Experimental): Stimulation at frontal sites with transcranial random noise stimulation (tRNS) to modulate frontal brain areas plasticity
  Interventions: Procedure: Frontal tRNS
- Sham/placebo tRNS (Sham Comparator): Transcranial random noise stimulation (tRNS) is applied only in the first and the last 30 seconds of the experimental procedure, thus resulting ineffective.
  Interventions: Procedure: Sham/placebo tRNS

INTERVENTIONS:
Procedure: Occipital tACS at IAF-2Hz — tACS applied to occipital areas at 2 Hz below the individual alpha frequency (IAF)
  Arms: Occipital tACS at IAF-2Hz
Procedure: Occipital tACS at IAF+2Hz — tACS applied to occipital areas at 2 Hz above the individual alpha frequency (IAF)
  Arms: Occipital tACS at IAF+2Hz
Procedure: Frontal tACS at 4-7 Hz — tACS applied to frontal areas at 4-7 Hz
  Arms: Frontal tACS at 4-7 Hz
Procedure: Occipital tRNS — tRNS applied to occipital brain regions
  Arms: Occipital tRNS
Procedure: Frontal tRNS — tRNS applied to frontal brain regions
  Arms: Frontal tRNS
Procedure: Sham/placebo tACS — tACS is activated only for 30 seconds and then turned off, thus resulting ineffective
  Arms: Sham/placebo tACS
Procedure: Sham/placebo tRNS — tRNS is activated only for 30 seconds and then turned off, thus resulting ineffective
  Arms: Sham/placebo tRNS

SUMMARY:
The hypothesis of the study is to investigate how different trm (tES) methods (transcranial Alternating Current Stimulation, tACS, and transcranial Random Noise Stimulation, tRNS) applied at different stimulation frequencies and networks can modulate the predictive mechanisms in human perception and cognition. This is an interventional, monocentric, cross-sectional randomized, single-blinded study on healthy adult volunteers, recruited through online advertisements, flyers and oral transmission. Volunteers will be recruited from the general population of young adults.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18-35 years.
* Normal or corrected to normal vision, as per anamnestic investigation.

Exclusion Criteria:

* Participants with a diagnosis of epilepsy (as per anamnestic investigation).
* Participants with major neurological disorders (as per anamnestic investigation).
* Participants that are currently under psychopharmacological treatment with tricyclic antidepressants (as per anamnestic investigation).
* Participants with metal implants in the brain, pacemakers, brain stimulators, cochlear implants (as per anamnestic investigation).

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-06-13 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral measures | During the procedure
  To study if tACS or tRNS delivered in different brain networks can modulate the learning of statistical regularities in the context of visual perception we will evaluate the following behavioral measures recorded in a computerized visual perception task: hit rate, miss, false alarms, correct rejections. These behavioral measures will allow to derive measures of sensitivity (d') and response criterion (Beta and C), according to the theoretical framework of the Signal Detection Theory (SDT).

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No